CLINICAL TRIAL: NCT01688557
Title: Prospective Randomised Trial Comparing New Technologies of Endoscopic Bowel Visualisation With Conventional Colonoscopy.
Brief Title: Trial on Innovative Technologies in Colonoscopy
Acronym: RCT-IC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Collaborators: Specialist Diagnostic and Therapeutic Center MEDICINA (Unknown)
Responsible Party: Principal Investigator, Miroslaw Szura, Assisstant Professor, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Innovations in colonoscopy
Record Dates: First submitted 2012-09-16; First posted 2012-09-20 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Polyps; Neoplasms; Inflammatory Bowel Disease
Keywords: narrow band imaging; dual focus; responsive insertion technique; scope guide; colonoscopy; colorectal cancer screening
MeSH Terms: conditions — Polyps; Neoplasms; Inflammatory Bowel Diseases | interventions — Narrow Band Imaging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Innovative colonoscopy (Experimental): Innovative colonoscopy performed using narrow band imaging and dual focus function (NBI + Dual Focus).
  Interventions: Device: Innovative colonoscopy (Olympus CF-HQ190F, NBI + Dual Focus)
- Conventional colonoscopy (Active Comparator): Conventional colonoscopy performed without innovative techniques assessed in this study.
  Interventions: Device: Conventional colonoscopy (Olympus CF-H180DL)

INTERVENTIONS:
Device: Innovative colonoscopy (Olympus CF-HQ190F, NBI + Dual Focus) — NBI and Dual Focus options will be used to classify lesions according to Sano and Kudo classifications.
  Arms: Innovative colonoscopy
Device: Conventional colonoscopy (Olympus CF-H180DL) — Conventional colonoscopy performed without innovative techniques used in experimental arm.
  Arms: Conventional colonoscopy

SUMMARY:
The trial will compare results of screening colonoscopy performed by means of conventional colonoscopy and using new visualisation techniques during endoscopic examination.

* Electronic colonoscopes Olympus CF-HQ190F with following options: magnetic positioning (Scope Guide), responsive insertion technology (RIT), dual focus function, narrow band imaging (NBI) will be used for innovative colonoscopies
* Electronic colonoscopes Olympus CF-H180DL with Scope Guide and NBI options will be used for conventional colonoscopies Endoscopists will archive all images and establish presumptive diagnosis based on the results of different visualisation techniques. All endoscopes will be attached to Olympus Evis Exera III system. Biopsy of all pathological lesions will be performed to establish final diagnosis. The main outcome measure is diagnostic accuracy of innovative colonoscopy in comparison with conventional technique.

DETAILED DESCRIPTION:
A total of 600 consecutive patients undergoing screening unsedated colonoscopy will be randomly assigned to innovative or conventional examination. Randomization will be based on computer-generated randomization lists. All patients will be blinded so they will not know which techniques will be used to assess lesions found in colon. In innovative colonoscopy group narrow band imaging (NBI) and Dual Focus (DF) function will be used to identify and classify all lesions acc. to Sano and Kudo classification. Endoscopic biopsy will be taken from all lesion and endoscopic diagnosis will be compared with final histological diagnosis. Thus sensitivity, specificity, diagnostic accuracy, predictive values, likelihood ratio and Youden index will be calculated. As secondary endpoints total examination time, coecal intubation rate and pain intensity (VAS scale) will be established. This study will help to establish whether new technologies used during colonoscopy may improve diagnostic possibilities and whether they prolong examination time or lead to increase of pain intensity afterwards.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* no previous abdominal surgery
* no colonoscopy during last 10 years

Exclusion Criteria:

* age < 40 and > 65 years
* large bowel resection in history
* colonoscopy performed during last 10 years
* contraindications for general anaesthesia
* ASA > IV
* pregnancy
* confirmed neoplastic disease
* cirrhosis (Child B or C) or ascites
* immunosuppressive therapy or steroids intake
* malabsorption syndrome

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2012-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of innovative colonoscopy | 1 year
  Diagnostic accuracy of innovative techniques used during colonoscopy (narrow band imaging and double focus option) will be assessed using StatSoft Statistica 10.0 software. All lesions will be classified acc. to Sano and Kudo classification during colonoscopy and results will be compared with histologic examination.

SECONDARY OUTCOMES:
Total examination time | 8-20 minutes
  Time of the whole procedure (from insertion of the colonoscope to removing of the whole instrument) will be compared in conventional and innovative colonoscopy.
Coecal intubation time | 5-15 minutes
  Time from insertion of colonoscope to visualisation of the coecum - always confirmed by a snapshot.
Pain intensity (VAS scale) | 0-10
  Pain intensity will be assessed during and after each colonoscopy using the Visual Analogue Scale. It will be assessed immediately after colonoscopy, 15 min, 30 min, 1 hour and 2 hours after the procedure.

OTHER OUTCOMES:
Sensitivity of innovative colonoscopy | 1 year
  The sensitivity of innovative colonoscopy will be assessed (in percentages) using StatSoft Statistica 10.0 software.
Specificity of innovative colonoscopy | 1 year
  The specificity of innovative colonoscopy will be assessed (in percentages) using StatSoft Statistica 10.0 software.
Positive predictive Value (PPV) od innovative colonoscopy | 1 year
  The positive predicting value of innovative colonoscopy will be assessed using StatSoft Statistica 10.0 software.
Negative predicting value (NPV) of innovative colonoscopy | 1 year
  The negative predictive value (NPV) of innovative colonoscopy will be assessed using StatSoft Statistica 10.0 software.
Youden's index for innovative colonoscopy | 1 year
  The Youden's index of innovative colonoscopy will be assessed using StatSoft Statistica 10.0 software.
Diagnostic odds ratio (DOR) for innovative colonoscopy | 1 year
  The diagnostic odds ratio (DOR) of innovative colonoscopy will be assessed using StatSoft Statistica 10.0 software.
Likelihood ratio for positive test results (LR+) | 1 year
  The likelihood ratio for positive test results of innovative colonoscopy will be assessed using StatSoft Statistica 10.0 software.
Likelihood ratio for negative test results (LR-) | 1 year
  The likelihood ratio for negative test results (LR-) of innovative colonoscopy will be assessed using StatSoft Statistica 10.0 software.
Area under the ROC curve (AUC) | 1 year
  Area under the ROC curve for innovative colonoscopy will be calculated using StatSoft Statistica 10.0 software.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslaw Szura, MD, PhD, Principal Investigator — I Department of General Surgery, Jagiellonian University; Radoslaw Pach, MD, PhD, Study Chair — I Department of General Surgery, Jagiellonian University
Locations (2):
- Poland (2):
  - Specialist Diagnostic and Therapeutic Center MEDICINA, Krakow, Malopolska
  - I Department of General Surgery, Jagiellonian University, Krakow, Malopolska

REFERENCES:
- [Result] Szura M, Pasternak A, Bucki K, Urbanczyk K, Matyja A. Two-stage optical system for colorectal polyp assessments. Surg Endosc. 2016 Jan;30(1):204-14. doi: 10.1007/s00464-015-4186-x. Epub 2015 Apr 4. PMID 25840894
- [Derived] Pasternak A, Szura M, Solecki R, Matyja M, Szczepanik A, Matyja A. Impact of responsive insertion technology (RIT) on reducing discomfort during colonoscopy: randomized clinical trial. Surg Endosc. 2017 May;31(5):2247-2254. doi: 10.1007/s00464-016-5226-x. Epub 2016 Sep 8. PMID 27631316
- [Derived] Szura M, Pasternak A, Solecki R, Matyja M, Szczepanik A, Matyja A. Accuracy of preoperative tumor localization in large bowel using 3D magnetic endoscopic imaging: randomized clinical trial. Surg Endosc. 2017 May;31(5):2089-2095. doi: 10.1007/s00464-016-5203-4. Epub 2016 Aug 29. PMID 27572063
- See also: The official site of the I Department of General Surgery, Jagiellonian University — http://www.rydygier.cm-uj.krakow.pl/
- See also: The official site of Specialist Diagnostic and Therapeutic Center MEDICINA — http://www.medicina.pl